CLINICAL TRIAL: NCT01874496
Title: Iron Absorption Mechanism From a Slow Release Iron Capsule Using the Gastric Delivery System
Brief Title: Iron Absorption From GDS Capsules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EK 2013-N-05
Record Dates: First submitted 2013-05-13; First posted 2013-06-11 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — Meals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- GDS, meal (Experimental): GDS, meal
  Interventions: Dietary Supplement: GDS, meal
- GDS, no meal (Experimental): GDS, no meal
  Interventions: Dietary Supplement: GDS, no meal
- control, no meal (Active Comparator): control, no meal
  Interventions: Dietary Supplement: control, no meal
- control, meal (Active Comparator): control, meal
  Interventions: Dietary Supplement: control, meal

INTERVENTIONS:
Dietary Supplement: GDS, no meal — GDS, no meal
  Arms: GDS, no meal
Dietary Supplement: GDS, meal — GDS, meal
  Arms: GDS, meal
Dietary Supplement: control, no meal — control, no meal
  Arms: control, no meal
Dietary Supplement: control, meal — control, meal
  Arms: control, meal

SUMMARY:
Slow release iron capsules have been designed based on the gastric delivery system. Iron absorption from those capsules administered with and without meals will be measured using stable iron isotopes.

ELIGIBILITY:
Inclusion Criteria:

* female,
* age 18-50 years,
* max. body weight 65 kg,
* serum ferritin < 35µg/l

Exclusion Criteria:

* pregnancy,
* lactation,
* regular intake of medication,
* blood donation or significant blood losses over the past 4 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
fractional iron absorption | 2, 4, 6, and 8 weeks

SECONDARY OUTCOMES:
serum isotope appearance | day 1, 15, 29 and 33

OTHER OUTCOMES:
Serum non transferrin bound iron | day 1, 15, 29 and 33

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Canton of Zurich, Switzerland